CLINICAL TRIAL: NCT01080807
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Tolerability of Armodafinil Treatment (150 mg) in Improving Clinical Condition Late in the Shift and in Improving Functional and Patient-Reported Outcomes in Adult Patients With Excessive Sleepiness Associated With Shift Work Disorder
Brief Title: Efficacy and Tolerability of Armodafinil in Adults With Excessive Sleepiness Associated With Shift Work Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cephalon (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C10953/4030
Record Dates: First submitted 2010-03-03; First posted 2010-03-04 (Estimated); Results first posted 2012-06-20 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-05

CONDITIONS: Excessive Sleepiness
MeSH Terms: conditions — Disorders of Excessive Somnolence | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 150 mg/day armodafinil (Experimental)
  Interventions: Drug: Armodafinil
- Matching placebo (Placebo Comparator)
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: Armodafinil — At the baseline visit, patients who continued to meet eligibility criteria were randomly assigned (1:1) to receive either 150 mg of armodafinil or matching placebo treatment only on nights worked for 6 weeks. Study drug was taken once nightly, 30 to 60 minutes prior to the start of the night shift, on nights worked. Armodafinil treatment was titrated as follows (only on nights worked): the first dose was 50 mg (1 tablet), the second and third doses were 100 mg (2 tablets), and the fourth and subsequent doses were 150 mg (3 tablets). Placebo tablets matching armodafinil tablets were administered on the same schedule.
  Other Names: R-modafinil; CEP-10953
  Arms: 150 mg/day armodafinil
Drug: Matching Placebo — At the baseline visit, patients who continued to meet eligibility criteria were randomly assigned (1:1) to receive either 150 mg of armodafinil or matching placebo treatment only on nights worked for 6 weeks. Study drug was taken once nightly, 30 to 60 minutes prior to the start of the night shift, on nights worked. Armodafinil treatment was titrated as follows (only on nights worked): the first dose was 50 mg (1 tablet), the second and third doses were 100 mg (2 tablets), and the fourth and subsequent doses were 150 mg (3 tablets). Placebo tablets matching armodafinil tablets were administered on the same schedule.
  Arms: Matching placebo

SUMMARY:
The primary objective of the study is to determine whether armodafinil treatment is more effective than placebo treatment in patients with excessive sleepiness associated with shift work disorder (SWD) by measuring improved clinical condition late in the shift, including the commute home.

ELIGIBILITY:
Inclusion Criteria:

1. The patient currently meets the criteria for Shift Work Disorder (SWD) for duration of at least 1 month.
2. The patient has the presence of excessive sleepiness late in the shift, including the commute home if applicable, with a Clinical Global Impression of Severity of Illness (CGI-S) rating of 4 or more at screening.
3. The patient has clinically significant difficulty in social or occupational functioning, with a Global Assessment of Function (GAF) score less than 70 (on clinician interview) at screening.
4. The patient has a Karolinska Sleepiness Scale (KSS) score of 6 or more at screening (visit 1) that is confirmed at baseline (visit 2).
5. The patient works at least 5 night shifts per month, of which at least 3 nights are consecutive, and plans to maintain this schedule.
6. The patient works night shifts or rotating shifts that include at least 6 hours between 2200 and 0800 (including the time period 0400 to 0800), and shifts are no longer than 12 hours in duration.
7. The patient is in good health, as judged by the investigator.
8. The patient is able to complete self-rating scales.
9. Women of childbearing potential (not surgically sterile or 2 years postmenopausal), must use a medically accepted method of contraception, and must continue use of 1 of these methods for the duration of the study (and for 30 days after participation in the study). Acceptable methods of contraception include: abstinence, barrier method with spermicide, steroidal contraceptive (oral, transdermal, implanted, and injected) in conjunction with a barrier method, or intrauterine device (IUD).
10. The patient is willing and able to comply with study restrictions and to attend regularly scheduled clinic visits as specified in this protocol

Exclusion Criteria:

1. The patient has mild or more severe obstructive sleep apnea (OSA) defined as an apnea/hypopnea index more than 5 as determined by daytime polysomnography (PSG).
2. The patient has a medical or psychiatric disorder causing clinically significant functional impairment or contributing to the patient's excessive sleepiness.
3. The patient is currently taking a medication or substance that is causing clinically significant functional impairment or contributing to the patient's excessive sleepiness.
4. The patient has a clinically significant treated or untreated medical condition.
5. The patient has a history of clinically significant suicidal ideation in the judgment of the principal investigator or is currently suicidal based on medical and psychiatric history.
6. The patient has a known hypersensitivity to armodafinil, racemic modafinil, or any component of the study drug tablets.
7. The patient has a history of any clinically significant cutaneous drug reaction, or a history of clinically significant hypersensitivity reaction, including multiple allergies or drug reactions.
8. The patient consumes caffeine including coffee, tea and/or other caffeine containing beverages or food averaging more than 600 mg of caffeine per day within 7 days of the baseline visit.
9. The patient uses any prescription or over-the-counter (OTC) drugs disallowed by the protocol within 30 days of the baseline visit.
10. The patient has been in a prior armodafinil study.
11. The patient has a history of alcohol, narcotic, or any other drug abuse.
12. The patient has a positive urine drug screen (UDS) without medical explanation at the screening visit.
13. The patient has a clinically significant deviation from normal on physical examination.
14. The patient is a pregnant or lactating woman.
15. The patient has used an investigational drug within 1 month of the screening visit.
16. The patient has a disorder that could interfere with the absorption, distribution, metabolism, or excretion of the investigational product.
17. The patient needs to use any of the excluded medications in this protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 385 (Actual)
Dates: Start 2010-03; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor's Medical Expert, Study Director — Cephalon
Locations (63):
- United States (63):
  - REM Medical Sleep Center, Phoenix, Arizona
  - REM Medical Clinical Research, Tucson, Arizona
  - Central Arkansas Research, Hot Springs, Arkansas
  - Clinical Study Centers LLC, Little Rock, Arkansas
  - Peninsula Sleep Center, Burlingame, California
  - Avastra Clinical Trials, Fountain Valley, California
  - Pacific Sleep Medicine Services Inc, Los Angeles, California
  - Southwestern Research Inc, Pasadena, California
  - Pacific Sleep Medicnie Services Inc, Redlands, California
  - Stanford University Medical Center, Redwood City, California
  - Dormir Clinical Trials, Inc., San Diego, California
  - Southwestern Research Inc, Santa Ana, California
  - St Johns Medical Plaza Sleep Disorders Center, Santa Monica, California
  - PAB Clinical Research, Brandon, Florida
  - MD Clinical, Hallandale, Florida
  - Compass Research LLC, Orlando, Florida
  - Broward Research Group, Pembroke Pines, Florida
  - Miami Research Associates, South Miami, Florida
  - Florida Sleep Institute, Spring Hill, Florida
  - Clinical Research Group of St Petersburg, St. Petersburg, Florida
  - SomnoMedics, Tampa, Florida
  - Neurotrials Research Inc, Atlanta, Georgia
  - Sleep Disorders Center of Georgia-Peachtree, Atlanta, Georgia
  - Sleep Disorders Center of Georgia-Gainesville, Gainesville, Georgia
  - Sleepmed Inc, Macon, Georgia
  - Chicago Research Center, Chicago, Illinois
  - Suburban Lung Associates, Elk Grove Village, Illinois
  - The Center for Sleep and Wake Disorders d/b/a Midwest Neuro, Danville, Indiana
  - Fort Wayne Neurological Center, Fort Wayne, Indiana
  - Rehabilitation Associates of Indiana, Indianapolis, Indiana
  - Goldpoint Clinical Research, Indianapolis, Indiana
  - University of Iowa Hospitals, Iowa City, Iowa
  - Vince and Associates Clinical Research, Overland Park, Kansas
  - Community Research, Crestview, Kentucky
  - Kentucky Research Group, Louisville, Kentucky
  - Helene A. Emsellem, MD, Chevy Chase, Maryland
  - Sleep Health Center, Brighton, Massachusetts
  - St Mary's of Michigan, Saginaw, Michigan
  - The Center for Sleep Medicine, Hattiesburg, Mississippi
  - Washington University Sleep Medicine Center, St Louis, Missouri
  - Clayton Sleep Institute LLC, St Louis, Missouri
  - Somnos Laboratories, Inc d/b/a Somnos Clinical Research, Lincoln, Nebraska
  - Clinical Research Center of Nevada, Las Vegas, Nevada
  - CliniLabs Inc, New York, New York
  - Duke Insomnia & Sleep Research Program, Durham, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - North Coast Clinical Trials Inc, Beachwood, Ohio
  - Community Research Inc, Cincinnati, Ohio
  - Tri State Sleep Disorders Center, Cincinnati, Ohio
  - North Star Medical Research LLC, Middleburg Heights, Ohio
  - Mercy St Anne Sleep Disorder Center, Toledo, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Southeastern PA Medical Institute, Broomall, Pennsylvania
  - Consolidated Clinical Trials, Jefferson Hills, Pennsylvania
  - CRI Worldwide, Philadelphia, Pennsylvania
  - Sleep Lab of Northeastern PA, Summit Hill, Pennsylvania
  - SleepMed of South Carolina, Columbia, South Carolina
  - Mid-South Neurology Center, Germantown, Tennessee
  - FutureSearch Trials of Neurology, Austin, Texas
  - Kingwood Research Institute, Kingwood, Texas
  - Sleep Therapy and Research Center, San Antonio, Texas
  - Avastra Clinical Trials, Midvale, Utah

REFERENCES:
- [Derived] Erman MK, Yang R, Seiden DJ. The effect of armodafinil on patient-reported functioning and quality of life in patients with excessive sleepiness associated with shift work disorder: a randomized, double-blind, placebo-controlled trial. Prim Care Companion CNS Disord. 2012;14(4):PCC.12m01345. doi: 10.4088/PCC.12m01345. Epub 2012 Aug 9. PMID 23251870
- [Derived] Erman MK, Seiden DJ, Yang R, Dammerman R. Efficacy and tolerability of armodafinil: effect on clinical condition late in the shift and overall functioning of patients with excessive sleepiness associated with shift work disorder. J Occup Environ Med. 2011 Dec;53(12):1460-5. doi: 10.1097/JOM.0b013e318237a17e. PMID 22104981

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 385 patients at 45 centers in the US met entry criteria and were considered eligible for enrollment into the study; 2 of these patients enrolled twice under different identification numbers. Of the 383 patients enrolled, 371 received at least 1 dose of study drug and were evaluated for safety; 12 patients withdrew before taking any study drug.
Pre-assignment Details: The study consisted of a 1- to 3-week screening period, a 1-week baseline period (followed by randomization), and a 6-week double-blind treatment period.
Groups:
- 150 mg/Day Armodafinil; Matching Placebo: At the baseline visit, patients who continued to meet eligibility criteria were randomly assigned (1:1) to receive either 150 mg of armodafinil or matching placebo treatment only on nights worked for 6 weeks. Study drug was taken once nightly, 30 to 60 minutes prior to the start of the night shift, on nights worked. Armodafinil treatment was titrated as follows (only on nights worked): the first dose was 50 mg (1 tablet), the second and third doses were 100 mg (2 tablets), and the fourth and subsequent doses were 150 mg (3 tablets). Placebo tablets matching armodafinil tablets were administered on the same schedule.
Period: Overall Study
Arm/Group | 150 mg/Day Armodafinil | Matching Placebo
Started | 193 (Nine patients randomly assigned to the armodafinil treatment group did not receive study drug.) | 190 (Three patients randomly assigned to the placebo treatment group did not receive study drug.)
Completed | 158 | 167
Not Completed | 35 | 23
Not completed — Adverse Event | 9 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Withdrawal by Subject | 7 | 2
Not completed — Protocol Violation | 7 | 6
Not completed — Lost to Follow-up | 6 | 4
Not completed — Noncompliance with drug administration | 1 | 1
Not completed — Noncompliance to study procedures | 1 | 1
Not completed — Began working day shift | 0 | 2
Not completed — Laid off or terminated from job | 1 | 2
Not completed — Stopped working consistent night shifts | 0 | 1
Not completed — Work schedule changing | 1 | 1
Not completed — Work schedule and travel | 0 | 1
Not completed — Switched to first shift | 1 | 0
Not completed — Moved away without notifying center | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 150 mg/Day Armodafinil | Matching Placebo | Total
Number analyzed (Participants) | 193 | 190 | 383
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 193 | 190 | 383
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 36.7 (10.71) | 36.1 (10.75) | 36.4 (10.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 90 | 175
  Male | 108 | 100 | 208
Region of Enrollment [Number; unit: participants]
  United States | 193 | 190 | 383

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With at Least Minimal Improvement From Baseline in the Clinical Global Impression of Change (CGI-C) Rating as Related to Late Shift Sleepiness at Endpoint
Description: The Clinical Global Impression of Change (CGI-C) is an assessment performed by the clinician, evaluating the change in the patient's symptoms over time. The clinician categorizes the change as: very much improved, much improved, minimally improved, no change, minimally worse, much worse, or very much worse. The data presented here represents the percentage of patients whose condition showed at least minimal improvement in the CGI-C rating as related to late shift sleepiness (defined as the period 0400-0800, including the commute home).
Time Frame: Baseline and week 6 (or last observation after baseline)
Population: The number of participants analyzed represents the number of participants with evaluable data.
Measure: Number; unit: Percentage of participants
Arm/Group | 150 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 177 | 182
Percentage of participants | 77 | 57

2. Secondary Outcome: Change From Baseline to Endpoint in Global Assessment of Function (GAF) Score
Description: The Global Assessment of Functioning (GAF) is a numeric scale (0 through 100) used by the clinician to rate the social, occupational, and psychological functioning of the patient. A higher score indicates superior functioning and fewer symptoms. The data presented here represents the mean change from baseline to endpoint in the GAF scores of each group.
Time Frame: Baseline and week 6 (or last observation after baseline)
Population: The number of participants analyzed represents the number of participants with evaluable data.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 177 | 182
Units on a scale | 9.4 (0.62) | 5.0 (0.64)

3. Secondary Outcome: Change From Baseline to Week 3 in Global Assessment of Functioning
Description: The Global Assessment of Functioning (GAF) is a numeric scale (0 through 100) used by the clinician to rate the social, occupational, and psychological functioning of the patient. A higher score indicates superior functioning and fewer symptoms. The data presented here represents the mean change from baseline in the GAF scores of each group.
Time Frame: Baseline and Week 3
Population: The number of participants analyzed represents the number of participants with evaluable data.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 168 | 175
Units on a scale | 6.9 (0.51) | 3.7 (0.52)

4. Secondary Outcome: Change From Baseline to Week 6 in Global Assessment of Functioning
Description: as for outcome 3
Time Frame: Baseline and Week 6
Population: The number of participants analyzed represents the number of participants with evaluable data.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 157 | 167
Units on a scale | 9.8 (0.66) | 4.9 (0.67)

5. Secondary Outcome: Change From Baseline to Endpoint in the Mean Karolinska Sleepiness Scale (KSS) Score
Description: The Karolinska sleepiness scale is a 10-point scale, on which the participant has to mark his sleepiness during the previous 10 minutes. The scale ranges from 1, which indicates "extremely alert", to 10, which indicates "extremely sleepy, can't stay awake". The KSS was performed by the participant at the baseline visit, week 3, and week 6 (or early termination visit). The score recorded is the average of 3 assessments within ±15 minutes at 0400, 0600, and 0800. The data presented here represents the mean change from baseline in the KSS scores of each group.
Time Frame: Baseline and week 6 (or last observation after baseline)
Population: The number of participants analyzed represents the number of participants with evaluable data.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 176 | 180
Units on a scale | -2.8 (0.16) | -1.8 (0.17)

6. Secondary Outcome: Change From Baseline to Week 3 in the Mean Karolinska Sleepiness Scale (KSS) Score
Description: as for outcome 5
Time Frame: Baseline and week 3
Population: The number of participants analyzed represents the number of participants with evaluable data.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 166 | 171
Units on a scale | -2.6 (0.16) | -1.6 (0.16)

7. Secondary Outcome: Change From Baseline to Week 6 in the Mean Karolinska Sleepiness Scale (KSS) Score
Description: as for outcome 5
Time Frame: Baseline and week 6
Population: The number of participants analyzed represents the number of participants with evaluable data.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 157 | 167
Units on a scale | -2.9 (0.17) | -1.8 (0.17)

8. Secondary Outcome: Percentage of Patients With at Least Minimal Improvement From Baseline in the Clinical Global Impression of Change (CGI-C) Rating as Related to Late Shift Sleepiness at Week 3
Description: as for outcome 1
Time Frame: Baseline and week 3
Population: Full analysis set defined as subjects who were assessed with CGI-C at baseline and at week 3
Measure: Number; unit: Percentage of participants
Arm/Group | 150 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 168 | 175
Percentage of participants | 78 | 51

9. Secondary Outcome: Percentage of Patients With at Least Minimal Improvement From Baseline in the Clinical Global Impression of Change (CGI-C) Rating as Related to Late Shift Sleepiness at Week 6
Description: as for outcome 1
Time Frame: Baseline and week 6
Population: Full analysis set defined as subjects who were assessed with CGI-C at baseline and at week 6
Measure: Number; unit: Percentage of participants
Arm/Group | 150 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 157 | 167
Percentage of participants | 80 | 56

10. Secondary Outcome: Change From Baseline to Endpoint in the Modified Sheehan Disability Scale (MSDS) Composite Score
Description: Mental-health related disability was assessed with the Modified Sheehan Disability Scale (MSDS). The MSDS has three 11-point items, and the participant is asked to rate, on a numerical scale, the extent to which emotional problems have disrupted her/his work, social life, and family life/home responsibilities over the last month. Each item is rated from 0, indicating "not at all", to 10, indicating "extremely". Scores for the items are summed for a possible score of 0 to 30. The MSDS was performed by the patient at the baseline visit, at Week 3, and at Week 6.
Time Frame: Baseline and week 6 (or last observation after baseline)
Population: Full analysis set defined as subjects who were assessed with MSDS at baseline and at Endpoint.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 176 | 181
Units on a scale | -6.6 (0.6) | -4.2 (0.62)

11. Secondary Outcome: Change From Baseline to Endpoint in the Modified Sheehan Disability Scale (MSDS) Work Item Score
Description: as for outcome 10
Time Frame: Baseline and week 6 (or last observation after baseline)
Population: Full analysis set defined as subjects who were assessed with MSDS at baseline and at Endpoint.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 176 | 181
Units on a scale | -2.2 (0.24) | -1.2 (0.25)

12. Secondary Outcome: Change From Baseline to Endpoint in the Modified Sheehan Disability Scale (MSDS) Social Life Item Score
Description: as for outcome 10
Time Frame: Baseline and week 6 (or last observation (or last observation after baseline))
Population: Full analysis set defined as subjects who were assessed with MSDS at baseline and at Endpoint.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 176 | 181
Units on a scale | -2.2 (0.23) | -1.5 (0.24)

13. Secondary Outcome: Change From Baseline to Endpoint in the Modified Sheehan Disability Scale (MSDS) Family Life Item Score
Description: as for outcome 10
Time Frame: Baseline and week 6 (or last observation after baseline)
Population: Full analysis set defined as subjects who were assessed with MSDS at baseline and at Endpoint.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 176 | 181
Units on a scale | -2.2 (0.23) | -1.5 (0.23)

14. Secondary Outcome: Change From Baseline to Endpoint in the Modified Sheehan Disability Scale (MSDS) Score - Days Missed Work or Unable to Carry Out Responsibilities
Description: as for outcome 10
Time Frame: Baseline and week 6 (or last observation after baseline)
Population: Full analysis set defined as subjects who were assessed with MSDS at baseline and at Endpoint.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 177 | 181
Units on a scale | -0.5 (0.10) | -0.4 (0.10)

15. Secondary Outcome: Change From Baseline to Endpoint in the Modified Sheehan Disability Scale (MSDS) Score - Number of Days of Reduced Productivity
Description: as for outcome 10
Time Frame: Baseline and week 6 (or last observation after baseline)
Population: Full analysis set defined as subjects who were assessed with MSDS at baseline and at Endpoint.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 177 | 181
Units on a scale | -1.4 (0.13) | -0.7 (0.14)

16. Secondary Outcome: Treatment Satisfaction Questionnaire for Medication (TSQM)- Effectiveness Score at Endpoint
Description: TSQM is a 14 question questionnaire assessing satisfaction with the medication. 4 scales are generated: side effects, effectiveness, convenience, and global satisfaction. Subjects responded to the questionnaire at Week 3, Week 6, and last observation after baseline. Optional responses are: Extremely Dissatisfied, Very Dissatisfied, Dissatisfied, Somewhat Satisfied, Satisfied, Very Satisfied, and Extremely Satisfied. From the responses, a scale score from 0 - 100 is calculated, with a higher score indicating greater satisfaction. Results from the Effectiveness scale are presented here.
Time Frame: Endpoint
Population: Full analysis set defined as subjects who completed the TSQM at Endpoint (Week 6 or last observation after baseline)
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 119 | 126
Units on a scale | 65.7 (2.46) | 46.1 (2.48)

17. Secondary Outcome: Treatment Satisfaction Questionnaire for Medication (TSQM)- Side Effects Score at Endpoint
Description: TSQM is a 14 question questionnaire assessing satisfaction with the medication. 4 scales are generated: side effects, effectiveness, convenience, and global satisfaction. Subjects responded to the questionnaire at Week 3, Week 6, and last post-baseline observation. Optional responses are: Extremely Dissatisfied, Very Dissatisfied, Dissatisfied, Somewhat Satisfied, Satisfied, Very Satisfied, and Extremely Satisfied. From the responses, a scale score from 0 - 100 is calculated, with a higher score indicating greater satisfaction. Results from the Side Effects scale are presented here.
Time Frame: Endpoint
Population: Full analysis set defined as subjects who completed the TSQM at Endpoint (Week 6 or last observation after baseline)
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 119 | 126
Units on a scale | 88.3 (1.62) | 96.3 (1.63)

18. Secondary Outcome: Treatment Satisfaction Questionnaire for Medication (TSQM)- Convenience Score at Endpoint
Description: TSQM is a 14 question questionnaire assessing satisfaction with the medication. 4 scales are generated: side effects, effectiveness, convenience, and global satisfaction. Subjects responded to the questionnaire at Week 3, Week 6, and last observation after baseline. Optional responses are: Extremely Dissatisfied, Very Dissatisfied, Dissatisfied, Somewhat Satisfied, Satisfied, Very Satisfied, and Extremely Satisfied. From the responses, a scale score from 0 - 100 is calculated, with a higher score indicating greater satisfaction. Results from the Convenience scale are presented here.
Time Frame: Endpoint
Population: Full analysis set defined as subjects who completed the TSQM at Endpoint (Week 6 or last observation after baseline)
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 119 | 126
Units on a scale | 82.5 (1.50) | 80.7 (1.51)

19. Secondary Outcome: Treatment Satisfaction Questionnaire for Medication (TSQM)- Global Satisfaction Score at Endpoint
Description: TSQM is a 14 question questionnaire assessing satisfaction with the medication. 4 scales are generated: side effects, effectiveness, convenience, and global satisfaction. Subjects responded to the questionnaire at Week 3, Week 6, and last observation after baseline. Optional responses are: Extremely Dissatisfied, Very Dissatisfied, Dissatisfied, Somewhat Satisfied, Satisfied, Very Satisfied, and Extremely Satisfied. From the responses, a scale score from 0 - 100 is calculated, with a higher score indicating greater satisfaction. Results from the Global Satisfaction scale are presented here.
Time Frame: Endpoint
Population: Full analysis set defined as subjects who completed the TSQM at Endpoint (Week 6 or last observation after baseline)
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 119 | 126
Units on a scale | 59.9 (2.72) | 44.1 (2.74)

20. Secondary Outcome: Change From Baseline to Endpoint in the Functional Outcomes of Sleep Questionnaire (FOSQ-10) Total Score
Description: FOSQ-10 consists of 10 questions, on a scale of 1-4(1=extreme difficulty 4=no difficulty), measures impact of sleepiness on activities of daily living. Lower score = more difficulty with activity due to lack of sleep. Total score = MEAN of subscale scores (vigilance, productivity, social outcome, intimacy, activity) multiplied by 5. Worst total score is 5 (maximum difficulty) the best is 20 (no difficulty). This data reports CHANGE in total score from baseline to endpoint, with higher (positive) values representing improvement. Worst possible CHANGE value would be -15 best would be +15.
Time Frame: Baseline and week 6 (or last observation after baseline)
Population: Full analysis set defined as subjects who were assessed with FOSQ-10 at baseline and at endpoint
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 174 | 177
Units on a scale | 3.3 (0.3) | 2.6 (0.32)

21. Secondary Outcome: Change From Baseline to Endpoint in the Functional Outcomes of Sleep Questionnaire (FOSQ-10) Activity Level Score
Description: FOSQ-10 consists of 10 questions rated on a scale of 1 to 4 (1=extreme difficulty and 4=no difficulty), and is used to measure the impact of daytime sleepiness on activities of daily living and quality of life. A total score and 5 subscale (vigilance, general productivity, social outcome, intimacy, and activity level) scores are calculated from the responses. Worst subscale score is 1 (maximum difficulty) and the best score is 4 (no difficulty). This score represents the CHANGE from Baseline in the Activity level subscale. Positive change scores represent improvement (possible range -3 to +3).
Time Frame: Baseline and week 6 (or last observation after baseline)
Population: Full analysis set defined as subjects who were assessed with FOSQ-10 at baseline and at endpoint
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 174 | 177
Units on a scale | 0.7 (0.07) | 0.5 (0.07)

22. Secondary Outcome: Change From Baseline to Endpoint in the Functional Outcomes of Sleep Questionnaire (FOSQ-10) General Productivity Score
Description: FOSQ-10 consists of 10 questions rated on a scale of 1-4 (1=extreme difficulty, 4=no difficulty), and is used to measure the impact of daytime sleepiness on activities of daily living and quality of life. A total score and 5 subscale (vigilance, general productivity, social outcome, intimacy, and activity level) scores are calculated from the responses. Worst subscale score is 1 (maximum difficulty) and the best score is 4 (no difficulty). This score represents the CHANGE from Baseline in the General Productivity subscale. Positive change scores represent improvement (possible range -3 to +3).
Time Frame: Baseline and week 6 (or last observation after baseline)
Population: Full analysis set defined as subjects who were assessed with FOSQ-10 at baseline and at endpoint
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 175 | 178
Units on a scale | 0.7 (0.07) | 0.6 (0.08)

23. Secondary Outcome: Change From Baseline to Endpoint in the Functional Outcomes of Sleep Questionnaire (FOSQ-10) Vigilance Score
Description: FOSQ-10 consists of 10 questions rated on a scale of 1-4 (1=extreme difficulty, 4=no difficulty), and is used to measure the impact of daytime sleepiness on activities of daily living and quality of life. A total score and 5 subscale (vigilance, general productivity, social outcome, intimacy, and activity level) scores are calculated from the responses. Worst subscale score is 1 (maximum difficulty) and the best score is 4 (no difficulty). This score represents the CHANGE from Baseline in the Vigilance subscale. Positive change scores represent improvement (possible range -3 to +3).
Time Frame: Baseline and week 6 (or last observation after baseline)
Population: Full analysis set defined as subjects who were assessed with FOSQ-10 at baseline and at endpoint
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 174 | 178
Units on a scale | 0.7 (0.07) | 0.5 (0.08)

24. Secondary Outcome: Change From Baseline to Endpoint in the Functional Outcomes of Sleep Questionnaire (FOSQ-10) Social Outcome
Description: FOSQ-10 consists of 10 questions rated on a scale of 1-4 (1=extreme difficulty, 4=no difficulty), and is used to measure the impact of daytime sleepiness on activities of daily living and quality of life. A total score and 5 subscale (vigilance, general productivity, social outcome, intimacy, and activity level) scores are calculated from the responses. Worst subscale score is 1 (maximum difficulty) and the best score is 4 (no difficulty). This score represents the CHANGE from Baseline in the Social Outcome subscale. Positive change scores represent improvement (possible range -3 to +3).
Time Frame: Baseline and week 6 (or last observation after baseline)
Population: Full analysis set defined as subjects who were assessed with FOSQ-10 at baseline and at endpoint
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 169 | 173
Units on a scale | 0.6 (0.09) | 0.5 (0.09)

25. Secondary Outcome: Change From Baseline to Endpoint in the Functional Outcomes of Sleep Questionnaire (FOSQ-10) Intimacy
Description: FOSQ-10 consists of 10 questions rated on a scale of 1-4 (1=extreme difficulty, 4=no difficulty), and is used to measure the impact of daytime sleepiness on activities of daily living and quality of life. A total score and 5 subscale (vigilance, general productivity, social outcome, intimacy, and activity level) scores are calculated from the responses. Worst subscale score is 1 (maximum difficulty) and the best score is 4 (no difficulty). This score represents the CHANGE from Baseline in the Intimacy subscale. Positive change scores represent improvement (possible range -3 to +3).
Time Frame: Baseline and week 6 (or last observation after baseline)
Population: Full analysis set defined as subjects who were assessed with FOSQ-10 at baseline and at endpoint
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 152 | 148
Units on a scale | 0.6 (0.08) | 0.5 (0.08)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded throughout the study, from screening through Week 6 (or early termination visit).
Arm/Group | 150 mg/Day Armodafinil | Matching Placebo
Serious Adverse Events (participants affected / at risk) | 0/184 | 1/187
Other Adverse Events (participants affected / at risk) | 55/184 | 22/187
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 150 mg/Day Armodafinil (N=184) | Matching Placebo (N=187)
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 150 mg/Day Armodafinil (N=184) | Matching Placebo (N=187)
Dry mouth (Gastrointestinal disorders) | 8 | 3
Headache (Nervous system disorders) | 28 | 13
Insomnia (Psychiatric disorders) | 12 | 3
Nausea (Gastrointestinal disorders) | 20 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days